CLINICAL TRIAL: NCT06079203
Title: ED-LEAD: Emergency Departments Leading the Transformation of Alzheimer's and Dementia Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-00516; U19AG078105-01A1 (NIH)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease Related Dementia; Alzheimer Disease
Keywords: Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- No intervention (No Intervention): No intervention, serving as a usual care control group
- Single intervention: Emergency Care Redesign (ECR) (Experimental)
  Interventions: Behavioral: Emergency Care Redesign (ECR)
- Single intervention: Nurse-led Telephonic Care (NLTC) (Experimental)
  Interventions: Behavioral: Nurse-led Telephonic Care (NLTC)
- Single intervention: Community Paramedic-led Transitions Intervention (CPTI) (Experimental)
  Interventions: Behavioral: Community Paramedic-led Transitions Intervention (CPTI)
- Two intervention: ECR and NLTC (Experimental)
  Interventions: Behavioral: Emergency Care Redesign (ECR); Behavioral: Nurse-led Telephonic Care (NLTC)
- Two interventions: ECR and CPTI (Experimental)
  Interventions: Behavioral: Emergency Care Redesign (ECR); Behavioral: Community Paramedic-led Transitions Intervention (CPTI)
- Two interventions: NLTC and CPTI (Experimental)
  Interventions: Behavioral: Nurse-led Telephonic Care (NLTC); Behavioral: Community Paramedic-led Transitions Intervention (CPTI)
- All interventions: ECR, NLTC, and CPTI (Experimental)
  Interventions: Behavioral: Emergency Care Redesign (ECR); Behavioral: Nurse-led Telephonic Care (NLTC); Behavioral: Community Paramedic-led Transitions Intervention (CPTI)

INTERVENTIONS:
Behavioral: Emergency Care Redesign (ECR) — Care Process Redesign: Care process redesign with a shared structured worksheet for data gathering, standardized assessment and referral. Education of all providers (Physician, Nurse, and Social Work Champion) on new processes at huddles and via on-line training, smart phone-compatible animated videos, faculty meetings, e-mail and from ED champions on shift
  CDS System: Alerts and new workflow to refer the dyad to social work or care manager. Continued use throughout study period and beyond
  Follow up: Within 72 hours of ED visit if discharged home Social Work Champion will have a single phone call. Triadic telephone encounter to ensure understanding of discharge plan, medication management and connection to community services
  Arms: All interventions: ECR, NLTC, and CPTI; Single intervention: Emergency Care Redesign (ECR); Two intervention: ECR and NLTC; Two interventions: ECR and CPTI
Behavioral: Nurse-led Telephonic Care (NLTC) — Telephonic support for dyad for safe ED to home care transition, and to enhance knowledge and management of AD/ADRD and co-morbid conditions. First call to dyad within 72 hours of index ED visit from Registered nurses. Each call ~30 minutes depending on needs and willingness of dyad. Calls also occur at 14 days, and at least monthly thereafter for 6 months. Dyad or nurse can initiate additional as-needed calls and coordinate care and care needs with other providers
  Arms: All interventions: ECR, NLTC, and CPTI; Single intervention: Nurse-led Telephonic Care (NLTC); Two intervention: ECR and NLTC; Two interventions: NLTC and CPTI
Behavioral: Community Paramedic-led Transitions Intervention (CPTI) — Community paramedics to provide coaching with dyad to improve medication management, outpatient follow up, understanding of red flags necessitating medical care. Home visit within ~5 days of index ED visit. One home visit and three telephone encounters over 30 days
  Arms: All interventions: ECR, NLTC, and CPTI; Single intervention: Community Paramedic-led Transitions Intervention (CPTI); Two interventions: ECR and CPTI; Two interventions: NLTC and CPTI

SUMMARY:
The purpose of this study is to improve the care of persons living with dementia (PLWD) and their informal care partners by addressing emergency and post-emergency care through different combinations of three PLWD-care partner dyad focused interventions. The primary aims are to use coaching to help connect PLWD and their care partners with community support and services to improve transitional care, quality of care, care satisfaction and reduce future ED visits and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* patients age 66 and older
* have at least one ICD-10 visit diagnoses for Alzheimer's Disease or Alzheimer's Disease Related Dementias (AD/ADRD) from an inpatient or outpatient encounter within the last 3 years of the ED visit and are discharged (observation patients included)

Exclusion Criteria:

* patients who are under 66 years old

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19200 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Emergency Department (ED) revisits | Up to 30 days

SECONDARY OUTCOMES:
Number of ED revisits | Up to 14 days
Number of ED revisits | Up to 6 months
Number of hospitalizations | Up to 14 days
Number of hospitalizations | Up to 30 days
Number of hospitalizations | Up to 6 months
Number of healthy days at home | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Since the outcomes data for this study is largely CMS data, the study team will not be able to share it. In fact, once the study ends, the study team won't be able to access the data. CMS data cannot be made available by the study team.